CLINICAL TRIAL: NCT04921007
Title: Analgesic Efficacy of Ultrasound Guided Sacral Erector Spinae Plane Block Versus Caudal Block in Pediatric Anorectal Surgery
Brief Title: Ultrasound Guided Sacral Erector Spinae Plane Block in Pediatric Anorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sameh Fathy (Other)
Responsible Party: Sponsor-Investigator, Sameh Fathy, Lecturer of anesthesia, ICU & pain management; Faculty of Medicine, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sacral ESP Block
Record Dates: First submitted 2021-06-03; First posted 2021-06-10 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Analgesia
Keywords: Erector spinae plane block; Ultrasound guided; Sacral; Anorectal surgery
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) Sacral ESP block (Active Comparator): Ultrasound guided sacral erector spinae plane (ESP) block will be performed in the lateral position under sterile conditions, and bupivacaine will be administered.
  Interventions: Procedure: Sacral ESP block; Drug: Bupivacaine Hydrochloride
- Group (B) Caudal block (Active Comparator): Ultrasound guided caudal block will be performed in the lateral position under sterile conditions, and bupivacaine will be administered.
  Interventions: Procedure: Caudal block; Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Procedure: Sacral ESP block — A high-frequency ultrasound linear probe covered with a sterile sheath will be placed longitudinally to the midline of the sacrum. The median sacral crests and erector spinae muscle will be visualized, then a 22-gauge, 50 mm needle will be advanced from cranial to caudal direction until its tip touch the sacral crest.
  Other Names: Ultrasound guided approach
  Arms: Group (A) Sacral ESP block
Procedure: Caudal block — A high-frequency ultrasound linear probe covered with a sterile sheath will be placed on to the sacrococcygeal region. The dura mater, epidural space, conus medullaris, sacral cornua, and sacrococcygeal ligament will be identified. Using the in-plane technique, a 22-gauge, 50 mm needle will be introduced to reach the sacral epidural space.
  Other Names: Ultrasound guided approach
  Arms: Group (B) Caudal block
Drug: Bupivacaine Hydrochloride — Following negative aspiration, a precalculated dose (0.5 ml/kg) of 0.25% bupivacaine will be injected.
  Other Names: Marcaine

SUMMARY:
This study will be conducted to evaluate efficacy of ultrasound guided sacral erector spinae plane block for postoperative analgesia in pediatric anorectal surgery in comparison to caudal block.

DETAILED DESCRIPTION:
Regional anesthesia in children has become increasingly popular over the past few decades. A variety of peripheral and central nerve blocks have been developed to ensure that perioperative pain can be effectively controlled. So, it possible to reduce the dose concentrations of systemic drugs and improved hemodynamic stability in high-risk patients. Erector spinae plane (ESP) block with various approaches been used in many surgeries and obtained great popularity despite of its novelty. After first description; lower thoracic, lumbar and sacral approaches were defined for postoperative analgesia. There are a few cases in which sacral ESP block was administered and reported.

The aim of this study is to compare postoperative analgesic effect of ultrasound guided sacral ESP block and caudal block. It is hypothesized that sacral ESP block will be comparable to caudal block as a promising effective alternative for analgesia in patients who will undergo pediatric anorectal surgery with fewer side effects.

This prospective, randomized, comparative clinical study will include 60 children who will be scheduled for elective anorectal surgery under general anesthesia in Mansoura university hospitals. Informed written consent will be obtained from parents of all subjects in the study after ensuring confidentiality. The study protocol will be explained to parents of all patients in the study who will be kept fasting prior to surgery. Patients will be randomly assigned to two equal groups (ESP and caudal) according to computer-generated table of random numbers using the permuted block randomization method. The collected data will be coded, processed, and analyzed using SPSS program. All data will be considered statistically significant if P value is ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) I and II patients.
* Scheduled for pediatric anorectal surgery

Exclusion Criteria:

* Parental refusal of consent.
* Children with developmental delays, mental or neurological disorders.
* Bleeding or coagulation diathesis.
* History of known sensitivity to the used anesthetics.
* Infection or redness at the injection site.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Duration for the first analgesic request | Up to 24 hours after the procedure
  The time of the first analgesic request for paracetamol in minutes will be recorded.

SECONDARY OUTCOMES:
Total analgesic requirements of paracetamol | Up to 24 hours after the procedure
  The amount of paracetamol consumption in milligrams given as a rescue analgesia
Improvement in pain scores | Up to 24 hours after the procedure
  Pain score from 0 to 10 (0 = no pain and 10 = the worst imaginable pain) is assessed postoperatively at 1, 2, 4, 8, 12, 24 hours
Changes in heart rate | Up to end of the surgery
  Heart rate (beat/min) is recorded at ten-minute intervals until the end of the surgery.
Changes in mean arterial blood pressure | Up to end of the surgery
  Blood pressure (mmHg) is recorded at ten-minute intervals until the end of the surgery.
Changes in postoperative emergence agitation scale | Up to 30 minutes after the procedure
  Agitation is assessed using the 5- step Cravero scale (1-5) every five minutes from awakening and for 30 minutes.(1:Obtunded with no response to stimulation, 2:Asleep but responsive to movement or stimulation, 3:Awake and responsive, 4:Crying, 5:Thrashing behaviour that requires restraint)
Value of parent satisfaction from the procedure | Up to 24 hours after the procedure
  The parents will be investigated postoperatively for the quality of the procedure verbally (0-10; 0=None, 10=total satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Sameh M El-Sherbiny, MD, Principal Investigator — Mansoura Faculty of Medicine
Locations (1):
- Department of Anesthesia, Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No